CLINICAL TRIAL: NCT05971199
Title: Phase II Study of Fruquintinib Combined With Sintilimab and TACE for Inoperable Primary Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Guoliang Shao, Head of Department of Interventional Therapy, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2021-385
Record Dates: First submitted 2023-07-10; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — HMPL-013; sintilimab

STUDY DESIGN:
Intervention Model Description: fruquintinib+sintilimab+TACE
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): Fruquintinib+sintilimab+TACE
  Interventions: Drug: Fruquintinib; Drug: Sintilimab; Device: Transcatheter arterial chemoembolization（TACE）

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib:5 mg capsule orally once daily on day 1-21 in 28-day cycles；
Drug: Sintilimab — Sintilimab: 200 mg i.v. every 3 weeks
Device: Transcatheter arterial chemoembolization（TACE） — Transcatheter arterial chemoembolization（TACE）

SUMMARY:
The goal of this prospective, interventional clinical trial is to evaluation of fruquintinib in combination with sintulimab and TACE for inoperable primary hepatocellular carcinoma for progression-free survival (PFS).

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the second most common cause of cancer death worldwide, accounting for approximately 745,000 deaths annually and 9.1% of all cancer-related deaths worldwide, with only about 30% of HCC patients having access to curative therapies. Most patients have intermediate to advanced disease and are usually treated with palliative therapy using TACE or systemic therapy (e.g., sorafenib, lenvatinib).

The efficacy of either sorafenib or lenvatinib as a single agent in the treatment of hepatocellular liver cancer remains limited, therefore, exploring combination therapy is one of the current research hotspots. A recent randomized, open, multicenter clinical study (TACTICS) enrolling patients with unresectable HCC showed that PFS was significantly prolonged to 25.2 months in the TACE combined with sorafenib treatment group, compared to 25.2 months in the TACE alone group. PFS was only 13.5 months in the TACE treatment group (HR=0. 59, 95%CI: 0.41-0. 87, P=0. 006). Median TTP was 24.1 months in the combination treatment group and 13.5 months in the TACE treatment group alone (HR=0. 56, 95%CL 0. 38-0. 83, P=0. 004).

Sintilimab, a recombinant fully human IgG4-type PD-1 monoclonal antibody, is an innovative drug developed by Sintilimab (Suzhou) Co. At the end of 2018, Sintilimab was officially approved by the NMPA of china for the treatment of relapsed or refractory classic Hodgkin's lymphoma (cHL) after at least second-line systemic chemotherapy. As a biosimilar to pembrolizumab, sintilimab has great potential to play a role similar to that played by pembrolizumab in primary hepatocellular carcinoma.

Fruquintinib is a potent small molecule VEGFR inhibitor developed by Hutchmed Ltd. with full intellectual property rights, with high kinase selectivity and inhibitory activity only for the VEGFR kinase family (VEGFR1, 2 and 3).On September 5, 2018, the NMPA of china officially approved fruquintinib for patients who have previously received fluorouracil-based, oxaliplatin and irinotecan-based chemotherapy, and for patients with metastatic colorectal cancer (mCRC) who have received prior or are not suitable for prior anti-vascular endothelial growth factor (VEGF) therapy, anti-epidermal growth factor receptor (EGFR) therapy (RAS wild type).

Therefore, based on previous studies, this study intended to select patients with unresectable primary hepatocellular carcinoma, and prospectively observe the efficacy and safety of fruquintinib in combination with sintilimab and TACE in the treatment of unresectable CNLC(China liver cancer staging) 2b-3a patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, male or female;
2. Patients diagnosed with primary hepatocellular carcinoma (HCC) based on clinical diagnosis or pathology;
3. Patients diagnosed with Chinese stage IIb-IIIa according to the Primary Liver Cancer Diagnostic and Treatment Protocol (2019 version), and evaluated by the investigator to be unable to undergo surgical treatment, such as resection, ablation or liver transplantation;
4. Imaging reports within 14 days prior to the intervention showed the presence of at least 1 target lesion measurable by CT or MRI, and the lesion is suitable for repeated accurate measurements;
5. Child-Pugh liver function rating: grade A or better B (≤7 points);
6. ECOG score: 0-1;
7. all lesions amenable to phase 1 or 2 (fractionated TACE) TACE therapy;
8. Good organ and bone marrow function. Blood count: WBC>4. 0 × 109/L, Hb>80g/L, PLT>75 ×109/L, NEUT>/ 1.5 × 109/L; coagulation function:International normalized (prothrombin time) ratio(INR) <1.2; liver function indexes: serum albumin (ALB) >3.5 g/dl, serum total bilirubin(TBIL) <1.5 times the upper limit of normal value (excluding biliary obstruction), serum transaminases (ALT and AST)<3 times the upper limit of normal value; renal function: serum myelin (CR) <1.5 times the upper limit of normal value;
9. Patients with positive hepatitis B surface antigen need to have received anti-hepatitis B treatment prior to inclusion in the study;
10. Signed an informed consent form, were compliant and cooperated with the follow-up.

Exclusion Criteria:

1. Hepatobiliary cell carcinoma, sarcomatoid hepatocellular carcinoma, mixed cell carcinoma and fibrous lamellar hepatocellular carcinoma;
2. With portal trunk or vena cava invasion;
3. Having received interventional treatment such as TACE within 2 years
4. Combined with medical contraindications that preclude any contrast-enhanced imaging (CT or MRI);
5. Previous systemic therapy;
6. Uncontrollable ascites, hepatic encephalopathy or bleeding esophagogastric fundic varices;
7. Hypertension that cannot be reduced to within normal limits with antihypertensive medication (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg);
8. Suffering from myocardial ischemia or myocardial infarction of grade II or higher, poorly controlled arrhythmia of grade II or higher myocardial ischemia or infarction, poorly controlled arrhythmia (QTc interval greater than or equal to 450 ms, QTc interval calculated in Fridericia metric).

   (calculated in Fridericia formula);
9. History of gastrointestinal bleeding within the past 3 months or a clear tendency of gastrointestinal bleeding, such as: esophageal varices at risk of bleeding, locally active ulcer lesions, fecal occult blood (++);
10. Pregnant or breastfeeding women; patients of childbearing potential who are unwilling or unable to use effective contraceptive measures
11. HIV-infected patients;
12. Those suspected of being allergic to the study drug;
13. Other circumstances that, in the judgment of the investigator, may affect the conduct of the clinical study and the determination of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2024-12-23 (Estimated); Study Completion 2024-12-23 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 1 year
  Progression free survival period refers to the period from the beginning of treatment to the time when patients with cancer progress is observed or death occurs for any reason.

SECONDARY OUTCOMES:
Object response rate(ORR) | Change from baseline tumor volume at 6 months
  The proportion of patients whose tumor volume reduction reaches the predetermined value and can maintain the minimum time limit. It is the sum of the proportion of complete response (CR) and partial response(PR).
Time to response(TTR) | through study completion, an average of 1 year
  Time to response
Disease control rate(DCR) | 1 year
  It is the sum of the proportion of complete response (CR), partial response(PR) and stable disease(SD).
Overall survival(OS) | 1 year
  (OS) is defined as the time from the patient's first dose of study drug until any cause of their death.
Time to progression(TTP) | 24 months
  Time from the beginning of treatment to the objective progression of tumor

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Shao, Principal Investigator — Zhejiang Cancer Hospital Hangzhou, Zhejiang, China
Locations (1):
- Guoliang Shao, Hangzhou, Zhejiang, China